

#### **Protocol B7451094**

# A RANDOMIZED, OPEN-LABEL, PARALLEL-GROUP STUDY TO EVALUATE THE SAFETY AND EFFICACY OF ABROCITINIB 100 MG AND 200 MG TABLETS IN PARTICIPANTS AGED 12 YEARS AND OLDER WITH MODERATE TO SEVERE ATOPIC DERMATITIS IN INDIA

Statistical Analysis Plan (SAP)

Version: 3

**Date:** 13 Jul 2023

PFIZER GENERAL BUSINESS



# **TABLE OF CONTENTS**

| LIST OF TABLES | 4 |
|------------------------------------------------------------------|----|
| LIST OF FIGURES | 4 |
| APPENDICES | 4 |
| 1. VERSION HISTORY | 5 |
| 2. INTRODUCTION | 6 |
| 2.1. Study Objectives, Endpoints, and Estimands | e |
| 2.1.1. Primary Estimand(s) | 7 |
| 2.1.2. Secondary Estimand(s) | 8 |
| 2.1.3. Additional Estimand(s) | 10 |
| 2.2. Study Design | 10 |
| 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS | 11 |
| 3.1. Primary Endpoint(s) | 11 |
| 3.2. Secondary Endpoint(s) | 12 |
| 3.2.1. Response based on IGA Score | 12 |
| 3.2.2. Response based on EASI-75 | 12 |
| 3.2.3. Response based on SCORAD75 | 12 |
| 3.2.4. Change from baseline in POEM Score | 12 |
| 3.2.5. Change from baseline in ADCT Score | 12 |
| 3.3. Other Endpoint(s) | 13 |
| 3.3.1. Incidence of Bone Safety Findings | 13 |
| 3.4. Baseline Variables | 13 |
| 3.5. Safety Endpoints | 13 |
| 3.5.1. Adverse Events | 13 |
| 3.5.2. Laboratory Data | 13 |
| 3.5.3. Vital Signs | 13 |
| 3.5.4. Electrocardiograms | 14 |
| 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS) | 14 |
| 5. GENERAL METHODOLOGY AND CONVENTIONS | 14 |

# PFIZER GENERAL BUSINESS



| 5.1. Hypotheses and Dec | eision Rules | 14 |
|---------------------------|--------------------------------------|----|
| 5.2. General Methods | | 14 |
| 5.2.1. Analyses for | Binary Endpoints | 14 |
| 5.2.2. Analyses for | Continuous Endpoints | 15 |
| 5.2.3. Analyses for | Categorical Endpoints | 15 |
| 5.3. Methods to Manage | Missing Data | 15 |
| 6. ANALYSES AND SUMMA | ARIES | 15 |
| 6.1. Primary Endpoint(s) | ) | 15 |
| 6.1.1. Incidence of | AEs/SAEs | 15 |
| 6.2. Secondary Endpoint | c(s) | 16 |
| 6.2.1. Response ba | sed on IGA Score | 16 |
| 6.2.2. Response ba | sed on EASI-75 | 16 |
| 6.2.3. Response ba | sed on SCORAD75 | 16 |
| 6.2.4. Change from | n baseline in POEM Score | 17 |
| 6.2.5. Change from | n baseline in ADCT Score | 17 |
| 6.3. Other Endpoint(s) | | 17 |
| 6.3.1. Incidence of | bone safety findings in knee MRI | 17 |
| 6.4. Subset Analyses | | 18 |
| 6.5. Baseline and Other S | Summaries and Analyses | 18 |
| 6.5.1. Baseline Sur | mmaries | 18 |
| 6.5.2. Study Condu | act and Participant Disposition | 18 |
| 6.5.3. Study Treatr | ment Exposure | 18 |
| 6.5.4. Concomitant | t Medications and Nondrug Treatments | 18 |
| 6.6. Safety Summaries an | nd Analyses | 18 |
| 6.6.1. Adverse Eve | ents | 18 |
| 6.6.2. Laboratory I | Data | 19 |
| 6.6.3. Vital Signs. | | 19 |
| 6.6.4. Electrocardio | ograms | 19 |
| 7 INTEDIM ANALYSES | | 10 |
| 7. INTERIM ANALTSES | | |

# PFIZER GENERAL BUSINESS



| 7.2. Inte | rim Analyses and Summaries | 19 |
|---|---|---|
| 8. APPENDIC | CES | 20 |
| | LIST OF TABLES | |
| Table 1. | Summary of Changes | 5 |
| Table 2. | Protocol-Required Safety Laboratory Assessments | 13 |
| Table 3. | Investigator's Global Assessment (IGA) Scores | 22 |
| Table 4. | Clinical Sign Severity Scoring Criteria for the Eczema Area and Severity Index (EASI) | 23 |
| Table 5. | Handprint Determination of Body Surface Area (BSA) | 24 |
| Table 6. | Eczema Area and Severity Index (EASI) Area Score Criteria | 24 |
| Table 7. | Eczema Area and Severity Index (EASI) Body Region Weighting. | 24 |
| Figure 1. | LIST OF FIGURES Study Design (Main Study) | 11 |
| | APPENDICES | |
| Appendix 1. S | ummary of Analyses | 20 |
| Appendix 2. I | Oata Derivation Details | 21 |
| Appendix 2.1. | Definition and Use of Visit Windows in Reporting | 21 |
| Appendix 2.2. | Investigator's Global Assessment (IGA) Scores | 21 |
| Appendix 2.3. | Eczema Area and Severity Index | 22 |
| Appendix 2.4. | Scoring Atopic Dermatitis | 25 |
| Appendix 2.5. | HSS Pedi-FABS | 26 |
| Appendix 3. L | ist of Abbreviations | 27 |
| Annendix 4 R | eferences | 28 |

# PFIZER GENERAL BUSINESS



# 1. VERSION HISTORY

 Table 1.
 Summary of Changes

| Version/<br>Date | Associated<br>Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| 1 | Original | N/A | N/A |
| 18 Feb 2022 | 21 Dec 2021 | | |
| 2<br>12 May 2022 | Amendment 1<br>23 Mar 2022 | Per India BoH's recommendation | Added SCORAD efficacy assessment for atopic dermatitis as a secondary endpoint. (Sections 2.1, 2.1.2, 3.2.3, 5.2.1, 6.2.3, Appendix 1, Appendix 2.4) |
| | | | Revised "abnormal developmental bone findings", "abnormal bone findings", "bone abnormalities" to "bone safety findings" in Sections 2.1, 2.1.3, 2.2, 3.3.1, 5.2.1, 6.3.1, Appendix 1. |
| | | | Removed text: "Photographic images of<br>the lesion will be taken as part of source<br>documentation, wherever possible." in<br>Appendix 2.2 and Appendix 2.3 to align<br>with Protocol Amendment 1. |
| | | | Added subset analysis based on monotherapy or combination therapy in Section 6.4. |
| 3<br>13 Jul 2023 | Amendment 1<br>23 Mar 2022 | Add safety population | Added safety population and details for FAS in the analysis sets in Section 4. |
| | | | Changed the analysis population from FAS to Safety in Sections 3.1, 6.1.1, 6.6 and Appendix 1. |
| | | | Removed 'randomized' in Sections 6.5.1 and 6.5.2 as tables will be summarized according to actual treatment. |

PFIZER GENERAL BUSINESS



#### 2. INTRODUCTION

This statistical analysis plan (SAP) provides the detailed methodology for summary and statistical analyses of the data collected in Study B7451094. This document may modify the plans outlined in the protocol; however, any major modifications of the primary endpoint definition or its analysis will also be reflected in a protocol amendment.

# 2.1. Study Objectives, Endpoints, and Estimands

| Objectives | Endpoints | Estimands |
|---|---|---|
| Primary: | Primary: | Primary: |
| To evaluate the safety of<br>abrocitinib in participants<br>aged 12 years and older<br>with moderate to severe<br>Atopic Dermatitis (AD) | • Incidence of adverse events (AEs) and serious adverse events (SAEs) | • The primary estimand for safety is the incidence of AEs and SAEs in participants aged 12 years and older with moderate to severe AD, from the time of first dose to Week 16, regardless of dosing compliance or treatment discontinuation. |
| Secondary: | Secondary: | Secondary: |
| To assess the efficacy of abrocitinib in participants aged 12 years and older with moderate to severe AD | <ul> <li>Response based on Investigator's Global Assessment (IGA) score of clear (0) or almost clear (1) and greater than or equal to 2 points improvement from baseline at Week 12</li> <li>Response based on achieving ≥75% improvement from baseline in the Eczema Area and Severity Index total score (EASI-75) at Week 12</li> <li>Response based on ≥75% improvement in Scoring Atopic Dermatitis total score (SCORAD75) at week 12</li> </ul> | • The secondary estimand is the treatment effect of abrocitinib on participants aged 12 years and older with moderate to severe AD, based on IGA response, EASI-75 response and SCORAD75 response from baseline to Week 12, considering patients who discontinued treatment as non-responders and based on outcome measures of POEM and ADCT from baseline to Week 12 and at all scheduled time points. Data collected after treatment discontinuation is excluded. |

PFIZER GENERAL BUSINESS



| | <ul> <li>Change from baseline in Patient-Oriented Eczema Measure (POEM) at Week 12 and at all scheduled time points</li> <li>Change from baseline in Atopic Dermatitis Control Tool (ADCT) at Week 12 and at all scheduled time points</li> </ul> | |
|---|---|---|
| Primary substudy | Primary substudy | <b>Primary substudy estimand(s):</b> |
| objective(s): | endpoints (as secondary | |
| | endpoints for B7451094): | |
| • To evaluate the potential | • The incidence of bone | • The primary substudy |
| effects of abrocitinib on | safety findings in knee | estimand is the incidence of |
| bone development in | MRI 1 year after | bone safety findings in knee |
| adolescent participants 12 | randomization in | MRI after 1 year of being |
| to <18 years of age, as | adolescent participants | exposed to abrocitinib in |
| 1 | | 1 |
| assessed by knee | exposed to abrocitinib | adolescent participants 12 to |
| assessed by knee<br>magnetic resonance | exposed to abrocitinib<br>100 mg and 200 mg once | adolescent participants 12 to <18 years of age, regardless of |
| 3 | <u> </u> | |

#### 2.1.1. Primary Estimand(s)

The primary estimand is the incidence of AE/SAE regardless of whether an intercurrent event occurs. The estimand is defined according to the primary objective and is in alignment with the primary endpoint. It includes the following 4 attributes:

- Population: Patients aged 12 years and older with moderate to severe AD, as defined by the inclusion and exclusion criteria, and who are randomized;
- Variable: Binary indicator of whether any AE/SAE occurred at least once;
- Intercurrent event(s): Dosing compliance or treatment discontinuation is not considered for analysis. All data collected (including data after discontinuation of treatment) are included.
- Population-level summary: Incidence rate of AEs/SAEs, defined as the number of participants with AEs/SAEs from the time of first dose to Week 16 divided by the number of participants, in each treatment arm.

# PFIZER GENERAL BUSINESS



#### 2.1.2. Secondary Estimand(s)

The secondary estimand 1 is the treatment effect of abrocitinib based on IGA response. This estimand is defined according to the secondary objective and in alignment with the secondary endpoint response based on IGA score. It includes the following 4 attributes:

- Population: Patients aged 12 years and older with moderate to severe AD, as defined by the inclusion and exclusion criteria, and who are randomized;
- Variable: Response based on IGA score of clear (0) or almost clear (1) and greater than or equal to 2 points improvement from baseline at Week 12; participants who discontinued intervention for any reason or required a rescue medication are considered as non-responders;
- Intercurrent event: The intercurrent event "intervention discontinuation for any reason" is addressed in the variable definition;
- Population-level summary: IGA response rate with 95% confidence interval (CI), in each treatment arm.

The secondary estimand 2 is the treatment effect of abrocitinib based on EASI-75 response. This estimand is defined according to the secondary objective and in alignment with the secondary endpoint response based on EASI-75. It includes the following 4 attributes:

- Population: Patients aged 12 years and older with moderate to severe AD, as defined by the inclusion and exclusion criteria, and who are randomized;
- Variable: Response based on improvement of ≥75% from baseline EASI score at Week 12; participants who discontinued intervention for any reason or required a rescue medication are considered as non-responders;
- Intercurrent event: The intercurrent event "intervention discontinuation for any reason" is addressed in the variable definition;
- Population-level summary: EASI-75 response rate with 95% CI, in each treatment arm.

The secondary estimand 3 is the treatment effect of abrocitinib based on SCORAD75 response. This estimand is defined according to the secondary objective and in alignment with the secondary endpoint response based on SCORAD75. It includes the following 4 attributes:

• Population: Patients aged 12 years and older with moderate to severe AD, as defined by the inclusion and exclusion criteria, and who are randomized;

PFIZER GENERAL BUSINESS



- Variable: Response based on improvement of ≥75% from baseline SCORAD total score at Week 12; participants who discontinued intervention for any reason or required a rescue medication are considered as non-responders;
- Intercurrent event: The intercurrent event "intervention discontinuation for any reason" is addressed in the variable definition;
- Population-level summary: SCORAD75 response rate with 95% CI, in each treatment arm.

The secondary estimand 4 is defined according to the secondary objective and in alignment with the secondary endpoint change from baseline in POEM scores. It includes the following 4 attributes:

- Population: Patients aged 12 years and older with moderate to severe AD, as defined by the inclusion and exclusion criteria, and who are randomized;
- Variable: Change from baseline in POEM scores at Week 12 and at all scheduled time points; data after treatment discontinuation or use of rescue medication at any time during the treatment period will be censored;
- Intercurrent event: The intercurrent event "intervention discontinuation for any reason" is addressed in the variable definition;
- Population-level summary: Mean and standard deviation (SD), in each treatment arm.

The secondary estimand 5 is defined according to the secondary objective and in alignment with the secondary endpoint change from baseline in ADCT scores. It includes the following 4 attributes:

- Population: Patients aged 12 years and older with moderate to severe AD, as defined by the inclusion and exclusion criteria, and who are randomized;
- Variable: Change from baseline in ADCT scores at Week 12 and at all scheduled time points; data after treatment discontinuation or use of rescue medication at any time during the treatment period will be censored;
- Intercurrent event: The intercurrent event "intervention discontinuation for any reason" is addressed in the variable definition;
- Population-level summary: Mean and SD, in each treatment arm.

#### PFIZER GENERAL BUSINESS



#### 2.1.3. Additional Estimand(s)

The primary substudy estimand is the incidence of bone safety findings in knee MRI after 1 year of being exposed to abrocitinib in adolescent participants 12 to <18 years of age, regardless of dosing compliance or treatment discontinuation. This estimand is defined according to the primary substudy objective and is in alignment with the primary substudy endpoint. It includes the following 4 attributes:

- Population: Patients aged 12 to <18 years with moderate to severe AD, as defined by the substudy inclusion and exclusion criteria;
- Variable: Binary indicator of whether the participant had bone safety findings in knee MRI 1 year after randomization;
- Intercurrent event(s): Dosing compliance or treatment discontinuation is not considered for analysis. All data collected (including data after discontinuation of treatment) are included.
- Population-level summary: Incidence rate of bone safety findings, defined as the number of participants with bone safety findings in knee MRI 1 year after randomization divided by the number of participants that received treatment during the substudy, in each treatment arm.

# 2.2. Study Design

This is a randomized, open-label, parallel-group study to evaluate the safety and efficacy of abrocitinib 100 mg QD and 200 mg QD tablets in participants aged 12 years and older with moderate to severe AD in India. There is a planned treatment duration of 12 weeks, with 4 weeks of off-treatment safety follow up thereafter. Study participants will be screened within 28 days prior to the first dose of investigational product to confirm that they meet the eligibility criteria for the study.

This study protocol also includes a substudy evaluating whether abrocitinib has any potential effects on adolescent bone with regard to bone safety findings in knee MRI. Adolescent participants (12 to < 18 years of age) will continue to receive investigational product until 1 year after randomization into the main study.

PFIZER GENERAL BUSINESS





Figure 1. Study Design (Main Study)

# 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS

#### 3.1. Primary Endpoint(s)

The primary endpoint is the incidence of AEs/SAEs, defined as the number of participants with treatment emergent adverse events, divided by the number of participants in the Safety Population (Section 4).

An adverse event will be considered treatment emergent relative to a given treatment if:

• The event starts on or after the first dose of study drug, but before the last dose plus the lag time of 28 days. The algorithm will not consider any events that started prior to the first dose date. If an AE starts on the same day as the first dose date, it will be considered treatment emergent.

or

The event was seen prior to the start of study drug but increased in severity during the effective duration of treatment.

#### PFIZER GENERAL BUSINESS



# 3.2. Secondary Endpoint(s)

# 3.2.1. Response based on IGA Score

The Investigator's Global Assessment of AD is scored on a 5-point scale (0-4), reflecting a global consideration of the erythema, induration and scaling (Appendix 2.2). Response is defined as a Week 12 score of clear (0) or almost clear (1), which also translates to a reduction of at least 2 points from baseline.

# 3.2.2. Response based on EASI-75

The EASI quantifies the severity of a subject's atopic dermatitis based on both severity of lesion clinical signs and the percent of body surface area (BSA) affected (Appendix 2.3). Response is defined as improvement of at least 75% from baseline in the EASI total score at Week 12.

# 3.2.3. Response based on SCORAD75

The SCORAD is a validated scoring index for AD, which combines extent (0-100), severity (0-18), and subjective symptoms (0-20) based on pruritus and sleep loss, each scored using a visual analog scale (0-10). The SCORAD total score for an individual ranges from 0 to 103 (Appendix 2.4). The extent score is set to missing if any of the body areas are missing. The severity score is set to missing if severity is missing for any of the subjective symptoms. The subjective symptom score is set to missing if either the itch score or the sleeplessness score is missing. The total score is set to missing if any of the 3 components is missing. Response is defined as improvement of at least 75% from baseline in the SCORAD total score at Week 12.

# 3.2.4. Change from baseline in POEM Score

The POEM is a validated 7-item patient-reported outcome (PRO) measure used to assess the impact of AD recalled over the past week. <sup>1-3</sup> Each item is scored from 0 (No days) to 4 (Every day). The POEM score is derived as the sum of scores from all 7 POEM items. The range of POEM score is 0 to 28, with higher scores indicating greater symptom burden. If one item is unanswered, this is scored as 0. If two or more items are unanswered, the POEM score is set to missing. Change from baseline in POEM score is derived for all scheduled time points. A positive mean change score indicates worsening of symptom burden over time.

# 3.2.5. Change from baseline in ADCT Score

The ADCT is a validated 6-item PRO measure used to assess patient-perceived AD control. <sup>4</sup>, <sup>5</sup> Each item is scored 0 to 4. The ADCT score is derived as the sum of scores from all 6 ADCT items. The range of ADCT score is 0 to 24, with higher scores indicating lower AD control. If one item is unanswered, the ADCT score is set to missing. Change from baseline in ADCT score is derived for all scheduled time points. A positive mean change score indicates worsening of AD control over time.

PFIZER GENERAL BUSINESS



#### 3.3. Other Endpoint(s)

The following additional endpoints will be derived for participants included in the substudy.

# 3.3.1. Incidence of Bone Safety Findings

The primary substudy endpoint is the incidence of bone safety findings in knee MRI after 1 year of being exposed to abrocitinib in adolescent participants 12 to <18 years of age. Bone safety findings will be adjudicated by the Safety Adjudication Committee.

#### 3.4. Baseline Variables

For all safety and efficacy analyses, baseline value is defined as the result of the last assessment performed prior to first dose of study treatment.

# 3.5. Safety Endpoints

# 3.5.1. Adverse Events

See Section 3.1.

# 3.5.2. Laboratory Data

Below is a list safety laboratory data that will be collected in the study. Change from baseline will be derived for laboratory parameters with scheduled post-baseline assessments.

Table 2. Protocol-Required Safety Laboratory Assessments

| Hematology | Chemistry | Lipid Profile <sup>a</sup> | Other |
|---|---|---|---|
| Hemoglobin | Urea | Total cholesterol | At screening only: |
| WBC count | sCr | LDL | • FSH <sup>b</sup> |
| Neutrophils (%, Abs) | sCysC (at Screening) | VLDL | Serum pregnancy test |
| Lymphocytes (%, Abs) | Estimated Creatinine | HDL | (β-hCG, for WOCBP |
| Platelets | Clearance | Triglycerides | only)c |
| Coagulation Panel | AST | | • HBsAg |
| (APTT, PT/INR) | ALT | | • HIV |
| | TBili | | • HCV |
| | Alkaline phosphatase | | • TB test (as per site |
| | | | standards) |

a. Fasting lipid profile panel require at least an 8 hour fast. If possible, participants should comply with fasting requirements at those visits detailed above.

#### 3.5.3. Vital Signs

Vital signs data include blood pressure and pulse rate.

#### PFIZER GENERAL BUSINESS

b. For confirmation of postmenopausal status only.

c. Urine pregnancy test (for WOCBP only) will be performed at all visits other than screening visits.



#### 3.5.4. Electrocardiograms

Electrocardiograms (ECG) parameters to be summarized include heart rate, PR, QT, QTcF and QRS.

# 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS)

| Population | Description |
|---|---|
| Enrolled | All participants who sign the informed consent document. |
| Full analysis set (FAS) | All participants randomly assigned to study intervention and who take at least 1 dose of study intervention. Participants will be analyzed according to the treatment arm they are randomized to. |
| Safety | All participants randomly assigned to study intervention and who take at least 1 dose of study intervention. Participants will be analyzed according to the treatment they actually received. |
| Substudy analysis set (SAS) | All participants who entered the substudy and who take at least 1 dose of study intervention during the substudy. |

For safety analyses, participants will be analyzed according to the treatment they actually received. On the other hand, for efficacy analyses, participants will be analyzed according to the treatment arm they are randomized to.

# 5. GENERAL METHODOLOGY AND CONVENTIONS

The study will be analyzed and reported once all randomized participants have completed all scheduled procedures (or discontinued) in the main study, i.e. at study participant data set release after the completion of the main study. The substudy will be analyzed and reported after the substudy data set release following last participant last visit in the substudy. The substudy report will include analyses that are discussed in Sections 6.1 (using the SAS), 6.3, 6.5, and Appendix 2.5.

# 5.1. Hypotheses and Decision Rules

This is a descriptive study, therefore there are no decision rules and statistical hypothesis testing to be performed. The objective of the study is to estimate safety and efficacy parameters, separately for each treatment arm.

# 5.2. General Methods

### 5.2.1. Analyses for Binary Endpoints

Binary endpoints (response based on IGA, EASI-75 and SCORAD75 and incidence of bone safety findings) will be presented using proportions together with the 95% confidence

PFIZER GENERAL BUSINESS



interval calculated using the normal approximation (or the Clopper-Pearson exact method when the estimated proportion is 0 or 1). Incidence of adverse events will be presented using frequency counts and percentages.

#### 5.2.2. Analyses for Continuous Endpoints

Continuous endpoints will be summarized using descriptive statistics, including the number of non-missing observations, mean, SD, median, first and third quartiles, minimum and maximum values. Descriptive summaries of the observed values and change from baseline for each time point will be provided, for each treatment arm.

# 5.2.3. Analyses for Categorical Endpoints

Categorical endpoints will be summarized by frequency counts and percentages. Unless otherwise specified, the calculation of percentages will include the missing category. Therefore, counts of missing observations will be included in the denominator and presented as a separate category.

# 5.3. Methods to Manage Missing Data

For the analysis of efficacy endpoints using descriptive statistics, missing values will not be imputed. For the analysis of safety endpoints, the sponsor data standard rules for imputation according to Clinical Data Interchange Standards Consortium (CDISC) and Pfizer Standards (CaPS) will be applied.

#### 6. ANALYSES AND SUMMARIES

# **6.1. Primary Endpoint(s)**

#### 6.1.1. Incidence of AEs/SAEs

- Estimand strategy: Treatment policy (Section 2.1.1).
- Analysis set: Safety (Section 4).
- Analysis methodology: Descriptive statistics.
- Intercurrent events and missing data: All adverse event data collected will be analyzed regardless of dosing compliance or treatment discontinuation; missing values will not be imputed.
- The number and proportion of participants who had treatment emergent adverse events will be presented for each treatment arm. Treatment emergent adverse events will be summarized according to type, frequency, severity, seriousness and relationship to abrocitinib in each treatment arm.

#### PFIZER GENERAL BUSINESS



# 6.2. Secondary Endpoint(s)

# **6.2.1.** Response based on IGA Score

- Estimand strategy: Composite (Section 2.1.2).
- Analysis set: FAS (Section 4).
- Analysis methodology: Descriptive statistics and 95% CIs.
- Intercurrent events and missing data: Missing data due to participant discontinuing treatment or from the study for any reason are considered non-response. In addition, participants who required a rescue medication are considered non-responders.
- The response rate along with the 95% CI will be estimated for each treatment arm. In addition, summary of IGA scores for all scheduled time points will be presented for each treatment arm.

#### 6.2.2. Response based on EASI-75

- Estimand strategy: Composite (Section 2.1.2).
- Analysis set: FAS (Section 4).
- Analysis methodology: Descriptive statistics and 95% CIs.
- Intercurrent events and missing data: Missing data due to participant discontinuing treatment or from the study for any reason are considered non-response. In addition, participants who required a rescue medication are considered non-responders.
- The response rate along with the 95% CI will be estimated for each treatment arm. In addition, summary of EASI scores for all scheduled time points will be presented for each treatment arm.

# 6.2.3. Response based on SCORAD75

- Estimand strategy: Composite (Section 2.1.2).
- Analysis set: FAS (Section 4).
- Analysis methodology: Descriptive statistics and 95% CIs.
- Intercurrent events and missing data: Missing data due to participant discontinuing treatment or from the study for any reason are considered non-response. In addition, participants who required a rescue medication are considered non-responders.

#### PFIZER GENERAL BUSINESS



• The response rate along with the 95% CI will be estimated for each treatment arm. In addition, summary of SCORAD total scores for all scheduled time points will be presented for each treatment arm.

# 6.2.4. Change from baseline in POEM Score

- Estimand strategy: While on treatment (Section 2.1.2).
- Analysis set: FAS (Section 4).
- Analysis methodology: Descriptive statistics.
- Intercurrent events and missing data: Data collected after treatment discontinuation or
  use of rescue medication at any time during the treatment period will be censored;
  missing values will not be imputed.
- Summary statistics for observed value and change from baseline in POEM Score will be presented for all scheduled time points, for each treatment arm.

# 6.2.5. Change from baseline in ADCT Score

- Estimand strategy: While on treatment (Section 2.1.2).
- Analysis set: FAS (Section 4).
- Analysis methodology: Descriptive statistics.
- Intercurrent events and missing data: Data collected after treatment discontinuation or use of rescue medication at any time during the treatment period will be censored; missing values will not be imputed.
- Summary statistics for observed value and change from baseline in ADCT Score will be presented for all scheduled time points, for each treatment arm.

# **6.3.** Other Endpoint(s)

# 6.3.1. Incidence of bone safety findings in knee MRI

- Estimand strategy: Treatment policy (Section 2.1.3).
- Analysis set: SAS (Section 4).
- Analysis methodology: Descriptive statistics and 95% CIs.
- Intercurrent events and missing data: All data collected will be analyzed regardless of dosing compliance or treatment discontinuation; missing values will not be imputed.

# PFIZER GENERAL BUSINESS



• The incidence rate of bone safety findings in knee MRI, along with the 95% CI will be estimated for baseline and End of Treatment (EOT) in the substudy, for each treatment arm. In addition, the types of bone safety findings will be summarized.

# 6.4. Subset Analyses

Summary statistics for the efficacy endpoints (Section 6.2) will be presented by subgroups according to whether the participants received monotherapy or combination therapy based on the permitted concomitant AD therapies in the protocol.

#### 6.5. Baseline and Other Summaries and Analyses

#### 6.5.1. Baseline Summaries

Demographic, baseline disesase characteristics, and medical history will be summarized by treatment arm according to CaPS.

#### 6.5.2. Study Conduct and Participant Disposition

Participants' evaluation, disposition, and discontinuation will be summarized by treatment arm according to CaPS.

# 6.5.3. Study Treatment Exposure

A summary of dosing compliance by treatment arm will be provided. Dosing compliance will be calculated as the percent of the number of doses of study drug the participant took out of the expected total number of doses. Number and percent of participants with compliance of <80 % and >120% will be provided for each treatment arm.

The exposure to study drug (computed as last dosing date – first dosing date + 1) will be summarized by treatment arm and according to duration categories (<1 week,  $\geq$ 1 week to <4 weeks,  $\geq$ 4 weeks to < 8 weeks,  $\geq$ 8 weeks to < 10 weeks, and  $\geq$ 10 weeks).

#### 6.5.4. Concomitant Medications and Nondrug Treatments

Prior drug and non-drug treatments, concomitant drug and non-drug treatments will be summarized for each treatment arm according to CaPS.

#### 6.6. Safety Summaries and Analyses

All safety analyses will be performed on the Safety population. These will be presented in a tabular format and summarized descriptively for each treatment arm following Pfizer standards as appropriate.

#### 6.6.1. Adverse Events

Medical Dictionary for Regulatory Activities (MedDRA) will be used to classify all AEs with respect to system organ class and preferred term. Summaries will include treatment

PFIZER GENERAL BUSINESS



emergent AEs/SAEs, withdrawal from active treatment due to AEs, and serious infections, defined as any infection (viral, bacterial, and fungal) requiring hospitalization or parenteral antimicrobials or meets other criteria that require it to be classified as a serious adverse event.

Any AEs that occur after signing Informed Consent and before randomization and the first dose of study drug will be listed but not summarized.

#### 6.6.2. Laboratory Data

Laboratory data will be listed and summarized according to CaPS. Laboratory parameters will be summarized descriptively at baseline, Week 4 and EOT visits, and will include the observed and change from baseline values.

### 6.6.3. Vital Signs

Vital signs will be summarized descriptively over time. Summaries will include the observed and change from baseline values. Height and weight will be summarized at baseline.

# 6.6.4. Electrocardiograms

ECG parameters will be summarized at baseline and EOT visits and will include the observed and change from baseline values.

# 7. INTERIM ANALYSES

#### 7.1. Introduction

No formal interim analysis will be conducted for this study. As this is an open-label study, the sponsor may conduct reviews of the data during the course of the study for the purpose of safety assessment. Interim safety and efficacy data after approximately 50% of the total sample size has been randomized in the study will be prepared and summarized to support presentation of initial results to India Bureau of Health (BoH). Additional summaries of interim data, including MRI data may be prepared to support presentation of results to regulatory agencies.

#### 7.2. Interim Analyses and Summaries

Data package to be provided to India BoH for presentation of initial results will include derived CDISC Study Data Tabulation Model (SDTM) datasets and data summaries that will include descriptive statistics of collected data on safety and efficacy parameters, as well as demographic and baseline characteristics.

PFIZER GENERAL BUSINESS



# 8. APPENDICES

# **Appendix 1. Summary of Analyses**

| Endpoint | Population | Data Inclusion and Rules for<br>Handling Intercurrent Events and<br>Missing Data | Analysis Method |
|---|---|---|---|
| Incidence of AEs/SAEs | Safety | All data collected will be included regardless of intercurrent events. Missing data will not be imputed. | Descriptive statistics |
| Response based on IGA<br>Score | FAS | Missing data due to discontinuation of treatment or from the study or use of rescue medication will be considered as non-response. | Descriptive statistics; point and interval estimation |
| Response based on EASI-75 | FAS | Missing data due to discontinuation of treatment or from the study or use of rescue medication will be considered as non-response. | Descriptive statistics; point and interval estimation |
| Response based on SCORAD75 | FAS | Missing data due to discontinuation of treatment or from the study or use of rescue medication will be considered as non-response. | Descriptive statistics; point and interval estimation |
| Change from baseline in POEM Score | FAS | Data collected after treatment discontinuation or use of rescue medication will be censored. Missing data will not be imputed. | Descriptive statistics |
| Change from baseline in ADCT Score | FAS | Data collected after treatment discontinuation or use of rescue medication will be censored. Missing data will not be imputed. | Descriptive statistics |

PFIZER GENERAL BUSINESS



| • | Substudy<br>Analysis<br>Set | All data collected will be included regardless of intercurrent events. Missing | Descriptive statistics; point and interval estimation |
|---|---|---|---|
| | | data will not be imputed. | estimation |

# **Appendix 2. Data Derivation Details**

# Appendix 2.1. Definition and Use of Visit Windows in Reporting

Visit windows will be used for efficacy variables.

| Visit Label | Target Day | Definition [Day window] |
|---|---|---|
| Baseline | Day 1 (Day of first | Last observation prior to and |
| | dose) | including day of first dose |
| Week 2 | 15 | Days 2 to 22 |
| Week 4 | 29 | Days 23 to 43 |
| Week 8 | 57 | Days 44 to 71 |
| Week 12 | 85 | Days 72 to 99 |
| Substudy EOT <sup>a</sup> | 366 | Days 353 to 380 or observation collected at Early Termination |
| Substudy Follow-up <sup>b</sup> | 394 | Days 381 to 408 or observation collected after Early Termination |

a. For MRI and HSS Pedi-FABS assessments in the Substudy

If two or more assessments fall into the same window, the assessment closest to the Target Day will be used. If two assessments are equally distant from the Target Day in absolute value, the later assessment will be used.

# Appendix 2.2. Investigator's Global Assessment (IGA) Scores

The Investigator's Global Assessment of AD is scored on a 5-point scale (0-4), reflecting a global consideration of the erythema, induration and scaling. The clinical evaluator of AD will perform an assessment of the overall severity of atopic dermatitis and assign an IGA

PFIZER GENERAL BUSINESS

b. For HSS Pedi-FABS assessments in the Substudy



score and category as described in Table 3. The assessment will be a static evaluation without regard to the score at a previous visit.

Table 3. Investigator's Global Assessment (IGA) Scores

| Score | Category | Description |
|---|---|---|
| 0 | Clear | Atopic dermatitis is cleared, except for any residual discoloration (post-inflammatory hyperpigmentation and/or hypopigmentation). |
| 1 | Almost Clear | Overall, the atopic dermatitis is not entirely cleared and remaining lesions are light pink (not including post inflammatory hyperpigmentation) and/or; have barely palpable hard thickened skin and/or papules and/or; have barely perceptible lichenification; excoriation and oozing/crusting are absent. |
| 2 | Mild | Overall, the atopic dermatitis consists of lesions that are light red; with slight, but definite hard thickened skin and/or papules; with slight, but definite linear or picked scratch marks or penetrating surface injury; with slight, but definite thickened skin, fine skin markings, and lichenoid scale; oozing/crusting is absent. |
| 3 | Moderate | Overall, the atopic dermatitis consists of lesions that are red; with easily palpable moderate hard thickened skin and/or papules; with moderate linear or picked scratch marks or penetrating surface injury; with moderate thickened skin, coarse skin markings, and coarse lichenoid scale; with slight oozing/crusting. |
| 4 | Severe | Overall, the atopic dermatitis consists of lesions that are deep, dark red; with severe hard thickened skin and/or papules; with severe linear or picked scratch marks or penetrating surface injury; with severe thickened skin with very coarse skin markings and lichenoid scale; with moderate to severe oozing/crusting. |

# **Appendix 2.3. Eczema Area and Severity Index**

The EASI quantifies the severity of a participant's AD based on both severity of lesion clinical signs and the percent of BSA affected. EASI is a composite scoring by the AD clinical evaluator of the degree of erythema, induration/papulation, excoriation, and lichenification (each scored separately) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body.

**Lesion Severity by Clinical Signs:** The basic characteristics of AD lesions - erythema, induration/papulation, excoriation, and lichenification-provide a means for assessing the PFIZER GENERAL BUSINESS



severity of lesions. Assessment of these four main clinical signs is performed separately for four body regions: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Average erythema, induration/papulation, excoriation, and lichenification are scored for each body region according to a 4-point scale: 0 = absent; 1 = mild; 2 = moderate; 3 = severe. Morphologic descriptors for each clinical sign severity score are shown in Table 4.

Table 4. Clinical Sign Severity Scoring Criteria for the Eczema Area and Severity Index (EASI)

| Score | | Description |
|---|---|---|
| Eryth | Erythema (E) | |
| 0 | Absent | None; may have residual discoloration (post-inflammatory |
| | | hyperpigmentation and/or hypopigmentation). |
| 1 | Mild | Light pink to light red |
| 2 | Moderate | Red |
| 3 | Severe | Deep, dark red |
| Indur | Induration/Papulation (I) | |
| 0 | Absent | None |
| 1 | Mild | Barely palpable to slight, but definite hard thickened skin and/or papules |
| 2 | Moderate | Easily palpable moderate hard thickened skin and/or papules |
| 3 | Severe | Severe hard thickened skin and/or papules |
| Excor | Excoriation (Ex) | |
| 0 | Absent | None |
| 1 | Mild | Slight, but definite linear or picked scratch marks or penetrating surface injury |
| 2 | Moderate | Moderate linear or picked scratch marks or penetrating surface injury |
| 3 | Severe | Severe linear or picked scratch marks or penetrating surface injury |
| Licher | Lichenification (L) | |
| 0 | Absent | None |
| 1 | Mild | Barely perceptible to slight, but definite thickened skin, fine skin markings, and lichenoid scale |
| 2 | Moderate | Moderate thickened skin, coarse skin markings, and coarse lichenoid scale |
| 3 | Severe | Severe thickened skin with very coarse skin markings and lichenoid scale |

**Percent BSA with Atopic Dermatitis:** The number of handprints of skin afflicted with AD in a body region can be used to determine the extent (%) to which a body region is involved

PFIZER GENERAL BUSINESS



with AD (Table 5). When measuring, the handprint unit refers to the size of each individual participant's hand with fingers in a closed position.

Table 5. Handprint Determination of Body Surface Area (BSA)

| Body Region | Total Number of<br>Handprints in Body<br>Region* | Surface Area of Body<br>Region Equivalent of One<br>Handprint* |
|---|---|---|
| Head and Neck | 10 | 10% |
| Upper Limbs | 20 | 5% |
| Trunk (including axillae and groin/genitals) | 30 | 3.33% |
| Lower Limbs (including buttocks) | 40 | 2.5% |

<sup>\*</sup>Handprint refers to the hand size of each individual participant.

The extent (%) to which each of the four body regions is involved with AD is categorized to a numerical Area Score using a non-linear scaling method according to the following BSA scoring criteria (Table 6).

Table 6. Eczema Area and Severity Index (EASI) Area Score Criteria

| Percent BSA with Atopic Dermatitis in a Body Region | Area Score |
|-----------------------------------------------------|------------|
| 0% | 0 |
| >0 - <10% | 1 |
| 10 - <30% | 2 |
| 30 - <50% | 3 |
| 50 - <70% | 4 |
| 70 - <90% | 5 |
| 90 - 100% | 6 |

**Body Region Weighting:** Each body region is weighted according to its approximate percentage of the whole body (Table 7).

Table 7. Eczema Area and Severity Index (EASI) Body Region Weighting

| Body Region | Body Region Weighting |
|----------------------------------|-----------------------|
| Head and Neck | 0.1 |
| Upper Limbs | 0.2 |
| Trunk (including axillae and | 0.3 |
| groin/genitals) | |
| Lower Limbs (including buttocks) | 0.4 |

PFIZER GENERAL BUSINESS



In each body region, the sum of the Clinical Signs Severity Scores for erythema, induration/papulation, excoriation, and lichenification is multiplied by the Area Score and by the Body Region Weighting to provide a body region value, which is then summed across all four body regions resulting in an EASI score as described in Equation 3.

```
Equation 3: EASI = 0.1Ah(Eh+Ih+Exh+Lh) + 0.2Au(Eu+Iu+ExU+Lu) + 0.3At(Et+It+Ext+Lt) + 0.4Al(El+Il+Exl+Ll)
```

A = Area Score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs

The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of AD.

The EASI Clinical Sign Severity Scores for each of the 4 body regions and the involvement by total number of handprints for each of the 4 body regions will be recorded on the CRF.

# **Appendix 2.4. Scoring Atopic Dermatitis**

SCORAD is a validated scoring index for atopic dermatitis, which combines extent (0-100), severity (0-18), and subjective symptoms (0-20) based on pruritus and sleep loss, each scored using a visual analog scale (0-10).

# Extent (A, maximum score of 100%)

To determine extent of AD, rule of 9 is used to calculate body surface area affected by AD as a percentage of the whole-body surface area. Body surface area as percentage of total body surface area for each body region is as follows:

- Head and neck 9%;
- Upper limbs 9% each;
- Lower limbs 18% each;
- Anterior trunk 18%;
- Back 18%;
- 1% for genitals.

The score for each body region is added up to determine the BSA affected by AD (A), which has a possible maximum score of 100%.

#### PFIZER GENERAL BUSINESS



# Severity (B, maximum score of 18)

A representative area of AD is selected. In this area, the severity of each of the following signs is assessed as none (0), mild (1), moderate (2) or severe (3).

- Erythema (reddening);
- Edema (swelling)/papulation;
- Oozing/crusting;
- Excoriation (scratch marks);
- Skin thickening (lichenification);
- Xerosis (dryness) (this is assessed in an area where there is no inflammation).

The severity scores are added together to give 'B' (maximum score of 18).

# Subjective Symptoms (C, maximum score of 20)

Subjective symptoms, ie, itch and sleep loss, are each scored by the participant or caregiver using a visual analog scale (VAS) where "0" is no itch (or no sleep loss) and "10" is the worst imaginable itch (or sleep loss). The value for each should reflect the average on a 10-point scale for the last 3 days/nights. These scores are added to give 'C' (maximum score of 20).

#### SCORAD Total Score

The SCORAD for an individual is calculated by the formula: A/5 + 7B/2 + C (can range from 0 to 103).

### Appendix 2.5. HSS Pedi-FABS

The Hospital for Special Surgery Pediatric Functional Activity Brief Scale (HSS Pedi-FABS) is a validated 8-item instrument designed to quantify the activity level of children between 10 and 18 years of age.<sup>6,7</sup> Two versions of the instrument based on the recall period will be implemented (1 month recall and 1 year recall). Items regarding running, cutting, decelerating, pivoting, duration, and endurance are scored 0 to 4, while items regarding completion and supervision are scored 0 to 3. The HSS Pedi-FABS score is derived as the sum of scores from all 8 items. The range of HSS Pedi-FABS score is 0 to 30, with higher

PFIZER GENERAL BUSINESS



scores indicating more physical activity. If one item is unanswered, the HSS Pedi-FABS score is set to missing.

Summary statistics for HSS Pedi-FABS score will be presented for all scheduled time points, for each treatment arm.

# **Appendix 3. List of Abbreviations**

| Abbreviation | Term |
|---|---|
| Abs | absolute |
| AD | Atopic Dermatitis |
| ADCT | Atopic Dermatitis Control Tool |
| AE | adverse event |
| ALT | alanine aminotransferase |
| APTT | Activated Partial Thromboplastin Time |
| AST | aspartate aminotransferase |
| β-hCG | beta-human chorionic gonadotropin |
| ВоН | Bureau of Health |
| BSA | body surface area |
| CaPS | CDISC and Pfizer Standards |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | confidence interval |
| CRF | Case Report Form |
| EASI | Eczema Area and Severity Index |
| EASI-75 | ≥75% improvement from baseline in the Eczema Area and Severity |
| | Index total score |
| ECG | Electrocardiogram |
| EOT | End of Treatment |
| FAS | Full analysis set |
| FSH | follicle-stimulating hormone |
| HBsAg | hepatitis B surface antigen |
| HCV | hepatitis C virus |
| HDL | high-density lipoprotein |
| HIV | human immunodeficiency virus |
| HSS Pedi-FABS | Hospital for Special Surgery Pediatric Functional Activity Brief |
| | Scale |
| IGA | Investigator's Global Assessment |
| INR | international normalized ratio |
| LDL | low-density lipoprotein |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | magnetic resonance imaging |
| POEM | Patient-Oriented Eczema Measure |

PFIZER GENERAL BUSINESS



| Abbreviation | Term |
|---|---|
| PR | pulse rate |
| PRO | patient-report outcome |
| PT | prothrombin time |
| QD | once daily |
| QTcF | corrected QT (Fridericia method) |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS | Substudy Analysis Set |
| SCORAD | SCORing Atopic Dermatitis |
| SCORAD75 | ≥75% improvement from baseline in the Scoring Atopic Dermatitis |
| | total score |
| sCr | serum creatinine |
| sCysC | serum Cystatin C |
| SD | standard deviation |
| SDTM | Study Data Tabulation Model |
| TB | tuberculosis |
| TBili | total bilirubin |
| VAS | Visual Analogue Scale |
| VLDL | very-low-density lipoprotein |
| WBC | white blood cell |
| WOCBP | woman/women of childbearing potential |

# **Appendix 4. References**

- 1. Charman C, Venn A, Williams HC. The Patient-Oriented Eczema Measure: development and initial validation of a new tool for measuring atopic eczema severity from the patients' perspective. Arch Dermatol 2004;140(12)(Dec):1513-9.
- 2. Charman CR, Venn AJ, Ravenscroft JC, et al.. Translating Patient-Oriented Eczema Measure (POEM) scores into clinical practice by suggesting severity strata derived using anchor-based methods. Br J Dermatol 2013;169(6)(Dec):1326-32.
- 3. Spuls PI, Gerbens LAA, Simpson E, et al. Patient-Oriented Eczema Measure (POEM), a core instrument to measure symptoms in clinical trials: a Harmonising Outcome Measures for Eczema (HOME) statement. Br J Dermatol 2017;176(4)(Apr):979-84.
- 4. Pariser DM, Simpson EL, Gadkari A, et al. Evaluating patient-perceived control of atopic dermatitis: design, validation, and scoring of the Atopic Dermatitis Control Tool (ADCT). Curr Med Res Opin. 2020;36(3):367-376.

PFIZER GENERAL BUSINESS



- 5. Simpson E, Eckert L, Gadkari A, et al. Validation of the Atopic Dermatitis Control Tool (ADCT©) using a longitudinal survey of biologic-treated patients with atopic dermatitis. BMC Dermatol. 2019 Nov 6;19(1):15.
- 6. Fabricant PD, Suryavanshi JR, Calcei JG, et al. The Hospital for Special Surgery Pediatric Functional Activity Brief Scale (HSS Pedi-FABS): Normative Data. Am J Sports Med. 2018 Apr;46(5):1228-34.
- 7. Fabricant PD, Robles A, Downey-Zayas T, et al. Development and Validation of a Pediatric Sports Activity Rating Scale: The Hospital for Special Surgery Pediatric Functional Activity Brief Scale (HSS Pedi-FABS). The American Journal of Sports Medicine. 2013;41(10):2421-9.

PFIZER GENERAL BUSINESS